CLINICAL TRIAL: NCT05643209
Title: Brugada Syndrome Substrate Characterization and Ablation: Insights From ECG BrS Type I Pattern, Novel Prognostic Index dST-Tiso and High Density Mapping
Brief Title: Brugada Syndrome Substrate Characterization and Ablation
Acronym: UNCOVERBrS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCH2022-02
Record Dates: First submitted 2022-11-17; First posted 2022-12-08 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- consecutive patients (Other): 20 patients clinically indicated for a endo-epicardial catheter-based mapping procedure for the treatment of ventricular tachycardia/ ventricular fibrillation substrate
  Interventions: Procedure: ablation

INTERVENTIONS:
Procedure: ablation — epicardial substrate homogenization (ablating abnormal fragmented prolonged low-frequency ventricular electrograms) in consecutive patients undergoing catheter ablation

SUMMARY:
Independent, single center, prospective study, to evaluate the efficacy, in consecutive BrS patients undergoing catheter ablation, at medium-long term follow-up after epicardial substrate homogenization. The target area is defined collecting signals using high density and high resolution mapping with equi-spaced electrode array. The ablation of abnormal fragmented prolonged low-frequency ventricular electrograms is performed by contact force catheter.

DETAILED DESCRIPTION:
Most of the patients with a diagnosis of Brugada syndrome (BrS) have no history of syncope or resuscitated cardiac arrest at the time of the diagnosis. Risk stratification in these patients is of utmost importance because cardiac arrest may be the presenting symptom. Individuals with a spontaneous electrocardiogram (ECG) BrS type I pattern (J-point and coved ST-segment elevation in the right precordial leads) are at higher risk of life-threating arrhythmic events than those with ECG abnormalities induced by sodium channel blocking agents. However, in the latter category, there may be subgroups of patients more exposed to the risk of arrhythmias. To date, a clear answer to this question has not yet emerged. Although controversial, programmed ventricular stimulation (PVS) is still central in the complex decision-making algorithm used to manage these lower risk BrS patients. A recent pooled analysis has confirmed the predictive role of PVS inidentifying BrS patients at increased risk of cardiac arrest6. Recently, Iacopino et al. demonstrate that the novel dST-Tiso interval >300 msec is a powerful predictor of ventricular arrhythmias inducibility (sensitivity 92% specificity 90%) in subjects with drug-induced BrS type I ECG pattern7. Radiofrequency ablation (RFA) of arrhythmogenic zones in the right ventricular epicardium has emerged over the past decade as a possible future curative treatment option for BrS. However, only a small number of studies with limited follow-up periods have reported successful results with RFA in symptomatic Brugada patients. The first to describe a successful RFA procedure in Brugada were Nademanee et al. using a selected cohort of nine high-risk patients with frequent ICD shocks for ventricular arrhythmias. More recently, Brugada et al.and Nademanee et al. described an improved technique for successful elimination of the Brugada syndrome phenotype with epicardial RFA. The mapping was performed before and after administration of flecainide/ajmaline which resulted in identification of more extensive arrhythmogenic segments in the RV epicardium beyond the RVOT.

Most recently, Iacopino et al. proposed a successful epicardial ablation of the arrhythmogenic substrate in BrS by using a novel and feasible technique with hybrid mini-thoracotomic approach and a 0-fluoroscopy strategy. The novel workflow combines both electrophysiological and surgical skills in a hybrid fashion with the aim to overcome their respective limitations.

Bipolar electrogram (BiEGM)-based substrate maps are heavily influenced by direction of a wavefront to the mapping bipole. Recently, Porta-Sanchez et al. evaluate high-resolution, orientation-independent peak-to-peak voltage (Vpp) maps obtained with an equi-spaced electrode array and omnipolar EGMs (OTEGMs), measure its beat-to-beat consistency, and assess its ability to delineate diseased areas within the myocardium compared against traditional BiEGMs on two orientations: along (AL) and across (AC) array splines and demonstrate that an equi-spaced electrode grid when combined with omnipolar methodology yielded the largest detectable bipolar-like voltage and is void of directional influences, providing reliable voltage assessment within infarcted and non-infarcted regions of the heart.

To date, there is no study that characterized the arrhythmogenic substrate of Brugada patients with the equi-spaced electrode array and omnipolar EGMs (OTEGMs) that are available nowadays.

The published studies regarding epicardial substrate ablation in Brugada patients describe an electrophysiological substrate characterized by abnormal fragmented prolonged low-frequency ventricular electrograms. We believe that the low resolution and the greater electrode dimensions of the conventional catheter can impact on both the duration and morphology of these signals.

The purpose of this study is to investigate the acute and long term efficacy of the protocol proposed which consists in ablating the abnormal fragmented prolonged low-frequency ventricular electrograms detected by equi-spaced electrode array and omnipolar EGMs (OTEGMs). Collecting and analyzing data concerning: late potential and voltage maps using different settings, vector data and speed maps, could be useful to better understand and describe the mechanism of this pathology.

In our expectation, a better definition of the abnormal substrate area dimension, could also confirm a relationship with the novel dST-Tiso interval.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic patients diagnosed with BrS-ECG pattern of types 1 and 2, both spontaneous and arising after Ajmaline tests, already implanted with an ICD.

   Symptomatic patients are defined as those who present ≥1 documented episode of VT / VF in the 12 months prior to enrollment.
2. Patients eligible for ablation with 3D high-density mapping system in accordance with national guidelines, IFU and according to medical decision;
3. Adult patients able to provide written informed consent

Exclusion Criteria:

1. Patients unable to provide written informed consent;
2. Patients unable to guarantee their presence at future FU visits;
3. Patients who, according to medical judgment, have a life expectancy of less than 12 months;
4. Patients who have undergone cardiac ablation in the 90 days prior to enrollment.
5. Patients who have had adverse events that have not been resolved after any invasive procedure;
6. Women potentially pregnant or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients free from any clinical ventricular arrhythmia at a 3, 6-months and 12-months follow-up from the procedure. | 12-months
  The primary aim of the study is the rate of success at medium-long term follow-up after epicardial substrate homogenization (ablating abnormal fragmented prolonged low-frequency ventricular electrograms) in consecutive brugada patients undergoing catheter ablation.
  The medium-long term success of the ablation is defined in terms of percentage of patients free from any clinical ventricular arrhythmia at a 3, 6-months and 12-months follow-up from the procedure.

SECONDARY OUTCOMES:
Collecting and analyzing data concerning late potential and voltage maps using different settings, vector data and speed maps, could be useful to better understand and describe the mechanism of this pathology. | 12 months
  • Comparison among different setting of voltage map (OT vs Standard acquisition)

CONTACTS AND LOCATIONS:
Overall Officials: Saverio Iacopino, MD, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iacopino S, Sorrenti PF, Petretta A, Colella J, Di Vilio A, Statuto G, Fabiano G, Campagna G, Peluso G, Fabiano E, Indellicati G, Brogneri S, Tremoli E, Mantovani L, Speziale G, Savini C, Tripodi A. Hybrid mini-thoracotomy for Brugada syndrome: epicardial substrate characterization and ablation-results from UNCOVER(BrS) study. Front Cardiovasc Med. 2025 Oct 28;12:1658355. doi: 10.3389/fcvm.2025.1658355. eCollection 2025. PMID 41229453